CLINICAL TRIAL: NCT02744508
Title: Comparison of Palonosetron Versus Combination of Palonosetron and Dexamethasone for Preventing Postoperative Vomiting in Patients Receiving Fentanyl by Patient-controlled Analgesia After Minor Orthopedic Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 4-2015-0232
Record Dates: First submitted 2016-04-18; First posted 2016-04-20 (Estimated); Last update posted 2018-06-20 (Actual); Status verified 2018-06

CONDITIONS: Orthopedic Surgery
Keywords: palonosetron, dexamethasone, PONV (postoperative nausea and vomiting)
MeSH Terms: conditions — Postoperative Nausea and Vomiting; Vomiting | interventions — Palonosetron; Dexamethasone

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- P group (Active Comparator): Palonosetron group
  Interventions: Drug: palonosetron
- PD group (Experimental): Palonosetron and dexamethasone group
  Interventions: Drug: palonosetron with dexamethasone

INTERVENTIONS:
Drug: palonosetron
  Arms: P group
Drug: palonosetron with dexamethasone
  Arms: PD group

SUMMARY:
Postoperative nausea and vomiting (PONV) is related with extended hospital day and risk factor of aspiration pneumonia. Postoperative patient controlled intravenous analgesia is related with postoperative nausea and vomiting. Selective 5-HT3 antagonist, Palonosetron, is the most recent medication for prevention of PONV. Purpose of our study is comparison of PONV preventive effect of palonosetron and combination of palonosetron and dexamethasone.

ELIGIBILITY:
Inclusion Criteria:

* patients who are undergoing minor orthopedic surgery.
* IV patient controlled analgesia

Exclusion Criteria:

* 1. minority (0~19 year)
* patients who are belongs to ASA class 3 or more, and have underlying complicated cardiovascular or psychological disease.
* Steroid medication
* Diabetes Mellitus medication

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 202 (Actual)
Dates: Start 2015-07-24 (Actual); Primary Completion 2017-03-20 (Actual); Study Completion 2017-03-20 (Actual)

PRIMARY OUTCOMES:
incidence of clinically significant PONV with PONV impact scale | 72 hours

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Anaesthesiology and Pain Medicine, Anaesthesia and Pain Research Institute, Yonsei University College of Medicine, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Myles PS, Weitkamp B, Jones K, Melick J, Hensen S. Validity and reliability of a postoperative quality of recovery score: the QoR-40. Br J Anaesth. 2000 Jan;84(1):11-5. doi: 10.1093/oxfordjournals.bja.a013366. PMID 10740540